CLINICAL TRIAL: NCT04693624
Title: Reproductive Outcome of IVF Treatment in Relation to the Early Luteal Phase Trajectory of Progesterone and Other Corpus Luteum Related Hormones
Brief Title: Early Luteal Hormones and IVF Outcomes After hCG Triggering
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 18/20/DD-BV
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Luteal Phase; in Vitro Fertilisation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hormonal levels: Blood samples are collected for analysis of progesterone, hCG, inhibin-A, and 17-OH-Progesterone levels.
  Interventions: Other: Hormonal levels

INTERVENTIONS:
Other: Hormonal levels — A total of ten (10) blood samples (2ml/each) will be collected during the study for subsequent analysis of progesterone, hCG, inhibin-A, and 17-OH-progesterone:
  Day of triggering (before the injection of hCG, appx. 6 pm) Twelve (12 hours) after hCG injection (appx. at 6 am) Twenty-four (24) hours after hCG injection (appx. at 6 pm) Thirty-six (36) hours after hCG injection (appx. at 8 am, 2 hours after OPU) One (1) day after OPU (60h after hCG) (appx. at 6 am) Two (2) days after OPU (84h after hCG) (appx. at 6 am) Three (3) days after OPU 108h after hCG) (appx. at 6 am) Four (4) days after OPU (132h after hCG) (appx. at 6 am) Five (5) days after OPU (156h after hCG) (appx. at 6 am) Six (6) days after OPU (180h after hCG) (appx. at 6 am)

SUMMARY:
It has recently been demonstrated that a bolus trigger of hCG induces various unphysiological conditions in the early luteal phase that may negatively affect an IVF treatment cycle's reproductive outcome. The bolus trigger of hCG differ from the natural cycle in mainly three different ways: 1) The timing of the initiation of hCG and progesterone rise is much faster after an hCG trigger than in the natural menstrual cycle 2) the maximal concentrations of hCG and progesterone considerably exceed those naturally observed 3) The timing of the peak progesterone concentration following an hCG trigger is advanced several days compared to the natural cycle. These characteristics may affect the reproductive outcome in treatment cycles but are not explored. The aim of this study is to monitor whether specific trajectories of important luteal phase hormones may predict the chances of conception?

DETAILED DESCRIPTION:
The early luteal phase after ovarian stimulation and final oocyte maturation using a bolus trigger of hCG is an area that has not received the same attention as regimes and protocols for ovarian stimulation during the follicular phase. The hCG trigger has been considered the golden standard since the beginning of the IVF era almost four decades ago. The hCG trigger serves two main functions: 1) it induces oocytes to advance meiosis to the metaphase of the second meiotic division ready for fertilization and further development, 2) secures stimulation of the corpora lutea to secrete progesterone (P4) during the early luteal phase due to its relatively long half-life. However, recent studies have suggested that each of these two functions may be optimized on their own and that better alternatives to the hCG trigger may be developed including a more physiological trigger for final maturation of follicles and individualized luteal phase support. However, only recently has the early luteal phase after IVF treatment using an hCG bolus trigger been described in studies involving more than just a few patients. These studies suggested that the unphysiological effects of the hCG trigger may be divided into three different categories: 1) The timing of the initiation of hCG and progesterone rise is much faster after an hCG trigger than in the natural menstrual cycle 2) the maximal concentrations of hCG and progesterone considerably exceed those naturally observed 3) The timing of the peak progesterone concentration following an hCG trigger is advanced several days compared to the natural cycle. How each of these effects influences pregnancy outcome in treatment cycles are currently unknown. Further, does characteristics shortly after administration of the hCG trigger for final oocyte maturation subsequently affect the reproductive outcome, and does this provide an opportunity for correcting or improving the luteal phase support given, with the improvement of clinical pregnancy rate as a result is also unknown. The aim of this study is to evaluate the trajectories of four hormones important for corpora lutea function (i.e. P4, 17-OH-P4, hCG, and inhibin-A) during the early luteal phase in women undergoing IVF treatment with luteal phase support given in the form of exogenous P4 administration and evaluate whether clinical pregnancy rates are related to specific characteristics of the early luteal phase. By including the measurements of 17-OH-P4 and inhibin-A the study will obtain an evaluation of the function of corpora lutea itself independent of the P4 administration provided.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 38
* BMI < 28kg/m2
* Normal ovarian reserve (anti-Müllerian hormone level above 8.93 pmol/L or an antral follicle count of 6 or above within two months prior to stimulation)
* Having 4 to 19 follicles with a diameter of 14mm or above on the day of hCG triggering
* Receiving a standard GnRH-antagonist protocol for ovarian stimulation
* Having indication for fresh embryo transfer
* Willingness to participate in the study, and to disclose any medical conditions to the investigator. The patient must be prepared and willing to comply with the requirements of the protocol.
* The patient should after appropriate oral and written consent understand the study and be informed that she may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Previous poor ovarian response (≤ 3 follicles) after appropriate FSH stimulation
* Hyper-response defined as ≥20 follicles ≥14 mm on the day of trigger
* Chronical medical conditions like Diabetes, Crohns disease, Thyroid disease, Hepatitis B, Sexually Transmitted Diseases and simultaneous participation in an interventional clinical trial.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Vietnamese women who will be indicated for IVF treatment with hCG administration for final oocytes maturation and undergo fresh embryo transfers.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate in relation to the trajectory of progesterone in the early luteal phase | After 24 weeks of gestation
  Live birth was defined as the birth of at least one newborn after 24 weeks' gestation that exhibited any sign of life (twins were a single count).
Live birth rate in relation to the trajectory of 17-OH progesterone in the early luteal phase | After 24 weeks of gestation
  Live birth was defined as the birth of at least one newborn after 24 weeks' gestation that exhibited any sign of life (twins were a single count).
Live birth rate in relation to the trajectory of hCG in the early luteal phase | After 24 weeks of gestation
  Live birth was defined as the birth of at least one newborn after 24 weeks' gestation that exhibited any sign of life (twins were a single count).

SECONDARY OUTCOMES:
The clinical pregnancy rate in relation to the trajectory of progesterone in the early luteal phase | At 5 weeks after embryo placement
  Pregnancy with at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity
The ongoing pregnancy rate in relation to the trajectory of progesterone in the early luteal phase | At 10 weeks or beyond after the embryo placement
  Pregnancy with detectable heart rate at 12 weeks' gestation or beyond
The clinical pregnancy rate in relation to the trajectory of 17-OH progesterone in the early luteal phase | At 5 weeks after embryo placement
  Pregnancy with at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity
The ongoing pregnancy rate in relation to the trajectory of 17-OH progesterone in the early luteal phase | At 10 weeks or beyond after the embryo placement
  Pregnancy with detectable heart rate at 12 weeks' gestation or beyond
The miscarriage rate in relation to the trajectory of progesterone in the early luteal phase | Before 12 weeks of gestation
  Pregnancy loss before 12 completed weeks of gestational age
The miscarriage rate in relation to the trajectory of 17-OH progesterone in the early luteal phase | Before 12 weeks of gestation
  Pregnancy loss before 12 completed weeks of gestational age
Live birth rate in relation to the trajectory of inhibin A in the early luteal phase | After 24 weeks of gestation
  Will be reported in a separate paper

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] N Vuong L, D Pham T, N A Ho V, T L Vu A, M Ho T, Yding Andersen C. In vitro fertilization outcome based on the detailed early luteal phase trajectory of hormones: a prospective cohort study. Reprod Biol Endocrinol. 2024 May 20;22(1):56. doi: 10.1186/s12958-024-01229-3. PMID 38769552